CLINICAL TRIAL: NCT00294632
Title: Lenalidomide and Rituximab Treatment of Relapsed Mantle Cell Lymphoma and Diffuse Large B-Cell Non-Hodgkin's Lymphoma, Transformed Large Cell Lymphoma, and/or Grade 3 Follicular Lymphoma (Follicular Cleaved Large Cell Lymphoma or Follicular Non-Cleaved Large Cell Lymphoma (RV-LYM-PI-0056)
Brief Title: Lenalidomide and Rituximab in the Treatment of Relapsed Mantle Cell Lymphoma (MCL) and Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0461; NCI-2012-01356 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Lymphoma
Keywords: Mantle Cell Lymphoma; B-Cell Non-Hodgkin's Lymphoma; Transformed Large Cell Lymphoma; Follicular Lymphoma; Lymphoma; MCL; Lenalidomide; CC-5013; Revlimid™; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell; Lymphoma, Follicular | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide + Rituximab (Experimental): Lenalidomide Starting Dose 10 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Starting Dose 10 mg By Mouth Daily on Days 1-21
  Other Names: CC-5013; Revlimid™
Drug: Rituximab — 375 mg/m^2 By Vein Weekly for 4 Weeks
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the drug lenalidomide (Revlimid, lenalidomide) that can be given with Rituxan® (rituximab) in the treatment of relapsed mantle cell lymphoma. The safety and effectiveness of this combination treatment will also be studied in both mantle cell lymphoma and diffuse large B-cell non-Hodgkin's lymphoma, transformed large cell lymphoma, and/or Grade 3 follicular lymphoma (follicular cleaved large cell lymphoma or follicular non-cleaved large cell lymphoma).

DETAILED DESCRIPTION:
Rituximab is a type of drug known as a monoclonal antibody. It is designed to act against the cluster of differentiation antigen 20 (CD20) antigen that is found on the surface of both normal B lymphocytes or on the malignant lymphoma cells. When rituximab attacks the CD20 antigen, it can kill the lymphoma cells. lenalidomide is known as an immunomodulatory drug. It is thought to work by helping the immune system fight disease.

If you are found to be eligible, you will receive lenalidomide plus rituximab. This study will be done in 2 phases. In the Phase I portion of this study, 6 dose levels of lenalidomide will be studied. The same level of rituximab will be given to all participants. Between 3-6 participants will be treated at each dose level. Those enrolled first on this study will receive the lowest dose of lenalidomide plus rituximab. After treatment, each dose level of lenalidomide will be evaluated to check for any intolerable side effects. The dose of lenalidomide that you will receive will depend on the time that you enter this study and the side effects of those participants that entered the study before you. Once a dose has been assigned to you, it will not increase, but it could decrease or remain the same for a while if you have intolerable side effects. Once the highest tolerable dose of lenalidomide has been found, additional participants will receive that dose during the Phase II portion of this study.

You should swallow lenalidomide capsules whole by mouth every day at the same time, with a glass of water on either a full or an empty stomach. Do not break, chew or open the capsules. This will continue for 21 days, followed by a 7-day rest period. Each 28-day period is called a cycle of therapy.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

During Cycle 1 only, you will also take rituximab by vein once a week for 4 weeks (total of 4 doses). The first rituximab infusion (by vein) usually takes 6 to 8 hours. Later infusions are generally shorter, taking about 4 hours to complete. For participants who have a large mass or who have lymphoma cells in their blood, the rituximab dose may be split into a 2-day infusion. Vital signs (temperature, blood pressure, respiration, and heart rate) will be monitored just before, during, and after the infusions. There will be an observation period of about 1 hour after the end of each rituximab infusion, after which you will be allowed to go home.

You will be given a diary to record when you take all of the study medications and any problems or illnesses you experience. You should also write down in the diary any other medications you take while you are on this study.

After you begin your treatment on the study drug, you will have check-up visits weekly for the first cycle, every 2 weeks for Cycles 2 and 3 of therapy, and then once a month for the rest of the study. If your doctor feels it is necessary, the check-up visits may take place more often. At the end of each 28-day treatment cycle, you will have a visit with the study doctor to see if it is safe for you to continue on this study and make sure the cancer has not gotten worse. If at the end of the each cycle, your doctor believes that you are eligible to continue (based on the degree and type of side effects you are having and the response of the cancer to the study drug), you will receive enough study drug for another 28-day treatment cycle.

At these visits you will have a complete physical exam, including measurement of vital signs. You will be asked questions about how you have felt since your last visit. All medications you have taken since your last visit will be reviewed by the study doctor. You should bring the empty pill packages and any unused medication along with the diary you were given earlier to each visit. You will have a blood sample collected (around 8 tablespoons) for routine blood tests to check on the status of the disease.

If you are eligible to continue on this study, a new 28-day supply of lenalidomide capsules will be given to you at this visit. Other tests may be done at these visits to check on the status of the disease. You may have a sample of bone marrow collected and/or have either x-rays or CT scans, positron emission tomography (PET) scan (if needed), and gastrointestinal endoscopy (for patients with known or suspected site of disease) to evaluate your response to therapy. These tests may not be done at every check-up visit. They will be done when your doctor feels they are necessary. You may have unscheduled visits at any time during this study if your doctor feels it is necessary for your care.

You may continue to receive treatment as long as the cancer does not get worse and you do not experience any intolerable side effects. If, at any time during treatment, the disease gets worse or you experience any intolerable side effects, you will be taken off this study, and your doctor will discuss other treatment options with you. The number of weeks you are on the study drug depends on how well you are tolerating the study drug and how well the lymphoma responds to the study drugs.

After your participation in this study ends, and if you have completed cycle 1 or more, you will have an end-of-study visit. At this visit you will have a complete physical exam, including measurement of vital signs and weight. You will have an ECG and you will be asked questions about how you have felt since your last visit. All medications you have taken since your last visit will be reviewed by the study doctor. You will have a blood sample collected (around 3 tablespoons) for routine blood tests to check on the status of the disease. You will have bone marrow collected for tests and have either x-rays or CT scans of your body to check on the status of the disease. You should return all empty drug packaging as well as any unused lenalidomide capsules at this visit.

If you completed at least 12 and no more than 24 cycles of treatment with lenalidomide, you will have follow-up visits every 3 months. If you complete 24 or more cycles of treatment with lenalidomide, you will have follow-up visits every 6 months. This will continue until the disease gets worse. At each visit, blood (about 1 teaspoon) will be drawn to test your thyroid function. The status of your disease will be evaluated and you may have a bone marrow biopsy and aspirate. You will have a chest x-ray and CT scans of the chest, abdomen, and pelvis. If needed, you will also have a CT scan of the neck. If needed, you will have a colonoscopy or endoscopy. You may also have a bone marrow biopsy and aspirate performed.

After the end-of-study visit, you will be contacted by phone every 6 months until March 15, 2015, to check on your health and for information about any other cancer treatments you may have received.

This is an investigational study. Lenalidomide is FDA approved and commercially available. Lenalidomide is approved for the treatment of patients with transfusion-dependent anemia due to Low- or Intermediate-1-risk myelodysplastic syndromes associated with the chromosome 5 abnormality with or without other chromosome abnormalities. Lenalidomide is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy. Its use in this study, for relapsed mantle cell lymphoma or large B-cell Non-Hodgkin's lymphoma, is investigational. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental.

Rituximab is FDA approved and commercially available for the treatment of non-Hodgkin's lymphomas.

Up to 71 participants with mantle cell lymphoma and 41 participants with diffuse large B-cell non-Hodgkin's lymphoma, transformed large cell lymphoma, and/or Grade 3 follicular lymphoma (follicular cleaved large cell lymphoma or follicular non-cleaved large cell lymphoma) will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I and Phase II: Confirmed diagnosis of mantle cell lymphoma with CD20 positivity in tissue biopsy. Patients must have previously treated relapsed and/or refractory MCL. Or for Phase II: Confirmed diagnosis of previously treated relapsed and/or refractory diffuse large B-cell lymphoma, transformed large cell lymphoma, and/or Grade 3 follicular lymphoma (follicular cleaved large cell lymphoma or follicular non-cleaved large cell lymphoma).
2. Understand and voluntarily sign an Institutional Review Board (IRB) approved informed consent form.
3. Age equal to or greater than 18 years at the time of signing the informed consent.
4. Patients must have bi-dimensional measurable disease (bone marrow only involvement is acceptable).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
6. Serum bilirubin <1.5 mg/dl and serum creatinine < 2.0 mg/dl; platelet count >75,000/mm^3 and absolute neutrophil count (ANC) > 1,000/mm^3. AST (SGOT) and ALT (SGPT) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present.
7. Disease free of prior malignancies of equal to or greater than 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years.
8. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test 10-14 days prior to therapy and repeated within 24 hours of starting study drug and must either commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide.
9. Continuation from # 8 : (HIGHLY EFFECTIVE METHODS - Intrauterine device (IUD), hormonal (birth control pills, injections, implants), tubal ligation, partner's vasectomy. ADDITIONAL EFFECTIVE METHOD-latex condom, diaphragm, cervical cap) while on study drug.
10. WCBP must agree to have pregnancy tests every week for the first 4 weeks of treatment, then every 4 weeks if her menstrual cycles are regular or every 2 weeks if her cycles are irregular, while on study drug, and 4 weeks after the last dose of study drug. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.
11. Patients may have 1 to 4 lines of prior therapy for MCL (projected median 2 prior lines of therapy). Patient may or may not have received an anthracycline-based chemotherapy regimen.
12. Patients must be willing to receive transfusions of blood products.
13. Past stem cell (autologous or allogenic) transplantation is acceptable.
14. Patients may have prior therapy with rituximab.

Exclusion Criteria:

1. Any serious medical condition including but not limited to, uncontrolled hypertension, diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active infection, active hemorrhage, laboratory abnormality, or psychiatric illness that places the patient at unacceptable risk and would prevent the subject from signing the informed consent form. Patients with history of cardiac arrythmias should have cardiac evaluation and clearance.
2. Pregnant or lactating females.
3. Use of any standard/experimental anti-lymphoma drug therapy, including steroids, within 3 weeks of initiation of the study or use of any experimental non-drug therapy (e.g., donor leukocyte/mononuclear cell infusions) within 56 days of initiation of the study drug treatment.
4. Known hypersensitivity to thalidomide or rituximab; including the development of erythema nodosum if characterized by a desquamating rash while taking thalidomide.
5. Prior use of lenalidomide.
6. Known HIV infection. Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; not including patients with positive serum Hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation.
7. All patients with history of central nervous system lymphoma.
8. Patients with peripheral blood involvement with white blood cell count (WBC) > 20,000 are EXCLUDED for the Phase I component of the study.
9. Patients with >/= Grade 3 neuropathy.
10. Patients with active pulmonary embolism or deep vein thrombosis (30 days within diagnosis).
11. Patients with severe bradycardia (heart rate <40 bpm, hypotension, light-headedness, syncope).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang M, Fayad L, Wagner-Bartak N, Zhang L, Hagemeister F, Neelapu SS, Samaniego F, McLaughlin P, Fanale M, Younes A, Cabanillas F, Fowler N, Newberry KJ, Sun L, Young KH, Champlin R, Kwak L, Feng L, Badillo M, Bejarano M, Hartig K, Chen W, Chen Y, Byrne C, Bell N, Zeldis J, Romaguera J. Lenalidomide in combination with rituximab for patients with relapsed or refractory mantle-cell lymphoma: a phase 1/2 clinical trial. Lancet Oncol. 2012 Jul;13(7):716-23. doi: 10.1016/S1470-2045(12)70200-0. Epub 2012 Jun 6. PMID 22677155
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 7, 2006 to February 21, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: There were 112 participants recruited for registration, 58 were screen failures prior to study inclusion
Groups:
- Phase I: Lenalidomide + Rituximab: Lenalidomide Starting Dose 10 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
- Phase II: Lenalidomide 20 mg + Rituximab: Lenalidomide MTD Dose 20 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
Period: Phase I Dose Escalation Period
Arm/Group | Phase I: Lenalidomide + Rituximab | Phase II: Lenalidomide 20 mg + Rituximab
Started | 14 | 0
Cohort 1: 10 mg | 3 | 0
Cohort 2: 15 mg | 3 | 0
Cohort 3: 20 mg | 6 | 0
Cohort 4: 25 mg | 2 | 0
Completed | 14 | 0
Not Completed | 0 | 0
Period: Phase II: 20 mg Lenalidomide
Arm/Group | Phase I: Lenalidomide + Rituximab | Phase II: Lenalidomide 20 mg + Rituximab
Started | 6 | 38
Completed | 6 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Lenalidomide + Rituximab: Lenalidomide Starting Dose 10 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Phase 1: Lenalidomide + Rituximab | Phase II: Lenalidomide 20 mg + Rituximab | Total
Number analyzed (Participants) | 14 | 38 | 52
Age, Continuous [Median (Full Range); unit: years] | 72 [56 to 84] | 64 [46 to 85] | 66 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 12 | 35 | 47
Region of Enrollment [Number; unit: participants]
  United States | 14 | 38 | 52

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide in Combination With Rituximab
Description: MTD is defined as the highest dose level in which 1 or fewer participants experienced a dose limiting toxicity (DLT) in 6 participants treated. DLT is any grade III or IV toxicity during the first 28 days (first cycle) of therapy.
Time Frame: 28 days of cycle 1
Measure: Number; unit: mg
Arm/Group | Phase I: Lenalidomide + Rituximab
Number analyzed (Participants) | 14
mg | 20

2. Secondary Outcome: Response of Participants Treated at Lenalidomide 20 mg
Description: Response definitions for measurable disease from the International Workshop Standardized Response Criteria for non-Hodgkin's Lymphoma: Complete Response (CR): Disappearance of all clinical evidence of active tumor for a minimum of four weeks. Partial Response (PR): =/>50% decrease in sum of products of all measured lesions persisting for >four weeks. No lesion may increase in size & no new lesion may appear. Minor Response (MR): >25% but less than 50% response. Stable Disease: Steady state or response less than minor & no progression for at least 8 weeks. There may be no appearance of significant new lesions. Progressive Disease: Unequivocal increase in size of any measurable lesion or appearance of significant new.
Time Frame: 56 days, assessed after 2 cycles
Population: Total analyzed includes Phase 2 participants (38) which includes six participants (6) that continued from Phase 1 who were treated with 20 mg Lenalidomide.
Measure: Count of Participants; unit: Participants
Groups:
- Lenalidomide 20 mg + Rituximab: Lenalidomide MTD Dose 20 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
Arm/Group | Lenalidomide 20 mg + Rituximab
Number analyzed (Participants) | 44
Participants
  Complete Response | 16
  Partial Response | 9
  Stable Disease | 10
  Progressive Disease | 9

3. Secondary Outcome: Objective Response Rate of Participants Treated With Lenalidomide 20 mg: Overall Response as % of Participants With Complete or Partial Response
Description: Objective response rate defined as percentage of participants with complete or partial response after 2 cycles of therapy maintained for one month. Objective response monitored using Simon's optimal 2-stage design.
Time Frame: 56 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 44
percentage of participants | 57

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of death from any cause or study completion, whichever came first, assessed up to 10 years
Description: Phase 1 included a total 14 participants in the MTD determination while Phase 2 included 38 additional participants, reflected in the Adverse Reporting are 6 participants from Phase I dosed at 20 mg MTD to total 44 participants in that portion of the study.
Groups:
- Phase I: Lenalidomide + Rituximab: Lenalidomide Starting Dose 10 mg, 15 mg, 20 mg or 25 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
- Phase II: Lenalidomide: Lenalidomide MTD Dose 20 mg oral daily on Days 1-21 + Rituximab 375 mg/m^2 intravenous weekly for 4 weeks
Arm/Group | Phase I: Lenalidomide + Rituximab | Phase II: Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/44
Serious Adverse Events (participants affected / at risk) | 9/14 | 24/44
Other Adverse Events (participants affected / at risk) | 14/14 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Lenalidomide + Rituximab (N=14) | Phase II: Lenalidomide (N=44)
Non-neutropenic infections (Infections and infestations) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 13 (13) — Grade 4 events
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) — Grade 4 events
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Grade 4 events
Thrombosis or thromboembolism (Vascular disorders) | 0 (0) | 1 (1) — Grade 4 events
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 0 (0) | 1 (1)
Altered mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 2 (3)
Snyocope (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Vascular disorders) | 1 (1) | 4 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Acute Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Post Radiation Treatment Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leucopenia/leukocytopenia (Investigations) | 1 (1) | 3 (3) — White blood cell decreased
Death (General disorders) | 1 (1) | 0 (0) — Unrelated, grade 4 non-neutropenic fever precursor
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Lenalidomide + Rituximab (N=14) | Phase II: Lenalidomide (N=44)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 38 (38)
Neutropenia (Blood and lymphatic system disorders) | 14 (14) | 44 (71)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14) | 42 (42)
Leucopenia (Blood and lymphatic system disorders) | 13 (13) | 44 (53)
Lymphopenia (Blood and lymphatic system disorders) | 14 (14) | 44 (64)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 22 (22)
Fatigue (General disorders) | 14 (14) | 38 (58)
Limb pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 19 (19)
Increased liver function (Investigations) | 11 (11) | 18 (18)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Non-neutropenic infections (General disorders) | 14 (14) | 28 (28)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (14) | 41 (41)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 30 (30)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (7) | 14 (14)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 30 (30)
Neuropathy (Nervous system disorders) | 0 (0) | 33 (33)
Nausea (Gastrointestinal disorders) | 0 (0) | 20 (20)
Vomiting (Gastrointestinal disorders) | 0 (0) | 15 (15)
Memory impairment (Nervous system disorders) | 0 (0) | 13 (13)
Mood alteration (Psychiatric disorders) | 0 (0) | 12 (12)
Dizziness (Nervous system disorders) | 0 (0) | 18 (18)
Blurred vision (Eye disorders) | 0 (0) | 15 (15)
Oral cavity pain (Gastrointestinal disorders) | 0 (0) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 23 (23)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 29 (29)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 29 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 8 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 14 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 15 (15)
Raised blood urea nitrogen (BUN) (Metabolism and nutrition disorders) | 0 (0) | 10 (10)
Raised Beta-2-Microglobulin (B2M) (Metabolism and nutrition disorders) | 0 (0) | 13 (13)
Raised Lactate dehydrogenase (LDH or LD) (Metabolism and nutrition disorders) | 0 (0) | 13 (13)
Facial oedema (General disorders) | 0 (0) | 4 (4)
Oedema limb (General disorders) | 0 (0) | 20 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 19 (19)
Red eyes (Eye disorders) | 0 (0) | 16 (16)
Thrombosis or thromboembolism (Hepatobiliary disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes